CLINICAL TRIAL: NCT05069636
Title: Lymphatic Osteopathic Manipulative Medicine to Enhance COVID-19 Vaccination Efficacy
Brief Title: Lymphatic Osteopathic Manipulative Medicine to Enhance Coronavirus (COVID-19) Vaccination Efficacy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The Principal Investigator left Rowan University School of Osteopathic Medicine.
Sponsor: Rowan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: PRO-2021-519
Record Dates: First submitted 2021-09-29; First posted 2021-10-06 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: COVID-19
Keywords: COVID-19; Osteopathic Manipulative Medicine; Antibody
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lymphatic OMM plus Moderna COVID-19 Vaccine regimen (Experimental): Patients receive OMM treatments that will include thoracic inlet and outlet myofascial release, pectoral traction myofascial release, and Miller Thoracic Lymphatic Pump technique plus the Moderna COVID-19 Vaccine regimen.
  Interventions: Other: Lymphatic OMM
- Light Touch plus Moderna COVID-19 Vaccine regimen (Sham Comparator): Patients receive a series of light touch techniques plus the Moderna COVID-19 Vaccine regimen.
  Interventions: Other: Light Touch

INTERVENTIONS:
Other: Lymphatic OMM — Patients receive lymphatic myofascial release and thoracic pump techniques.
  Arms: Lymphatic OMM plus Moderna COVID-19 Vaccine regimen
Other: Light Touch — Patients receive a series of light touch techniques.
  Arms: Light Touch plus Moderna COVID-19 Vaccine regimen

SUMMARY:
The purpose of this project is to study the impact of Osteopathic Manipulative Medicine (OMM) treatments, such as lymphatic myofascial release and thoracic pump techniques severe acute respiratory syndrome-associated coronavirus 2 (SARS-Cov-2) antibody levels in patients who receive the mRNA-1273 (Moderna) COVID-19 vaccine and to consider if these OMM strategies allow a stronger more robust immune response.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria will include age greater than 18 years old and having safely received the COVID-19 vaccine.

Exclusion Criteria:

* Exclusion criteria will include age under 18 years old, malignancy/cancer, ongoing infection, coagulopathy history, use of anticoagulant medications, and fracture or acute injury of the torso neck or upper extremities. Lymphatic OMM is safe during pregnancy and this does not need to be an exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-02-14 (Actual); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
severe acute respiratory syndrome-associated coronavirus 2 (SARS-Cov-2) antibody levels | The day of first vaccine dose (baseline), the day of second vaccine dose (at about 4-weeks post first vaccine dose), and 2-weeks post second vaccine dose (at about 6-weeks post first vaccine dose
  Antibody levels collected via blood draw

CONTACTS AND LOCATIONS:
Locations (1):
- Rowan University School of Osteopathic Medicine, Stratford, New Jersey, United States